CLINICAL TRIAL: NCT00662246
Title: A Phase I Dose Escalation Study Using Proton Beam Radiotherapy for Hepatocellular Carcinoma
Brief Title: Dose Escalation Study Using Proton Beam Radiotherapy for Hepatocellular Carcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Tae Hyun Kim, National Cancer Center Korea
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCCTS-07-225
Record Dates: First submitted 2008-04-10; First posted 2008-04-21 (Estimated); Last update posted 2012-04-03 (Estimated); Status verified 2012-03

CONDITIONS: Carcinoma, Hepatocellular
MeSH Terms: conditions — Carcinoma, Hepatocellular

ARMS (1):
- 1 (Experimental): Primary objectives :
  * to determine the recommended dose (i.e., the safest and most effective dose) by evaluating frequency of patients developing unacceptable (grade 3 or higher) acute toxicities attributable to proton beam radiotherapy for HCC.
  Interventions: Radiation: respiratory gated proton beam radiotherapy

INTERVENTIONS:
Radiation: respiratory gated proton beam radiotherapy — - Prescription dose to PTV as according to the following dose escalation schema: Dose level 1: 60 GyE /20 fx, 3GyE fraction dose, 5 days/week. Dose level 2: 66 GyE /22 fx, 3GyE fraction dose, 5 days/week. Dose level 3: 72 GyE /24 fx, 3GyE fraction dose, 5 days/week.

SUMMARY:
The radical treatment for Hepatocellular carcinoma (HCC) is surgery. However, it is only for 10 to 20% of all patients and 10 to 30% of them have relapsed every year after surgery. For an inoperable case, we can consider Liver transplantation. But there is not enough organ donor and it is very expensive. In that case, various treatment modalities for HCC (i.e., transcatheter arterial embolization [TAE] and percutaneous ethanol injection [PEI], radiofrequency ablation etc.) have become clinically available. In addition, after these treatment, radiation therapy can be conducted as a combined treatment. If it is difficult, radiation therapy can be conducted alone. In this case, radiation therapy can use fractionated stereotactic radiation therapy [FSRT] or 3D simulation to minimize the exposure to normal tissues. In recent years, Proton therapy is a new radiation therapy which remaining energy is released when they reach the tumor, delivering the most effective dose of radiation. The purpose of this trial is to improve the therapeutic effects by using proton therapy.

ELIGIBILITY:
Inclusion Criteria:

* HCC diagnosed as:

  * (i) the presence of risk factors including hepatitis B or C virus and liver cirrhosis, a serum a-fetoprotein (AFP) level greater than 400 IU/ml and a radiologically compatible feature with HCC in one or more CT/MRI/angiograms
  * (ii) the presence of risk factors including hepatitis B or C virus and liver cirrhosis, a serum a-fetoprotein (AFP) level less than 400 IU/ml, and a radiologically compatible feature with HCC in two or more CT/MRI/angiograms or (iii) histological confirmation
* HCC patients who were not prospective suitable or refused for any other treatment, such as surgery or local ablation therapy, or recurrent or residual tumor after other treatments.
* Without evidence of extrahepatic metastasis
* All target tumors must be encompassable within single irradiation field (12x12 cm maximum)
* No previous treatment to target tumors by other forms of RT
* Digestive tract not in contact with clinical target volume
* Liver function of Child-Pugh class A or B
* Age of ≥ 18 years
* Performance status of 0 to 2 on the Eastern Cooperative Oncology Group (ECOG) score
* WBC count ≥ 2,000/mm3; hemoglobin level ≥ 7.5 g/dL; platelet count ≥ 25,000/mm3; and adequate hepatic function (total bilirubin ≤ 3.0 mg/dL; AST and ALT < 5.0× upper limit of normal; no ascites)
* No serious comorbidities other than liver cirrhosis

Exclusion Criteria:

* Evidence of extrahepatic metastasis
* Age < 18 years
* Liver function of Child-Pugh class C
* Previous history of other forms of RT adjacent to target tumors
* Poor performance status of 3 to 4 on the Eastern Cooperative Oncology Group (ECOG) score
* Diffusely infiltrating tumor which is difficult to define the gross tumor volume accurately
* Multicentric HCCs, except for those with the following two conditions:

  * (i) multinodular aggregating HCC that could be encompassed by single clinical target volume and within single irradiation field (15x15 cm maximum)
  * (ii) lesions other than targeted tumor that were judged as controlled with prior surgery and/or local ablation therapy
* Digestive tract in contact with clinical target volume
* Pregnant or breast feeding status
* Previous history uncontrolled other malignancies within 2 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2007-01; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
all cause mortality | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Center Korea, Goyang-si, Gyeonggi-do, South Korea